CLINICAL TRIAL: NCT05514860
Title: The Impact of "First-Line" Rhythm Therapy on AF Progression
Acronym: PROGRESSIVE-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Jason Andrade, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H16-00617_SRG-15-P15-001
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoballoon-based PVI (Active Comparator): Sinus rhythm control via a pulmonary vein isolation (PVI) ("first-line") procedure utilizing the the Arctic Front Cryoballoon Procedure.
  Interventions: Procedure: Cryoballoon-based PVI
- Anti-Arrhythmic Drug Therapy (Active Comparator): Sinus rhythm control via the use of anti-arrhythmic drug (AAD) therapy ("first-line") based on local clinical practice, and according to guideline-suggested drug management for symptomatic patients with paroxysmal AF.
  Interventions: Drug: Anti-Arrhythmic Drug Therapy

INTERVENTIONS:
Procedure: Cryoballoon-based PVI — Patients randomized to first-line cryoballoon (CB) ablation will have the pulmonary vein isolation procedure performed according to standard clinical practice using the Arctic Front Cryoballoon ablation catheter. No anti-arrhythmic drugs will be prescribed in this arm.
  Arms: Cryoballoon-based PVI
Drug: Anti-Arrhythmic Drug Therapy — Antiarrhythmic drug therapy (Class I - flecainide, propafenone; Class III - sotalol, dronedarone) will prescribed and monitored based on local clinical practice, and according to guideline-suggested drug management for symptomatic patients with paroxysmal AF.
  Arms: Anti-Arrhythmic Drug Therapy

SUMMARY:
The PROGRESSIVE-AF Trial is a national, multi-center randomized controlled trial comparing early ("first-line") catheter-based pulmonary vein isolation (PVI) using cryothermal energy to first-line anti-arrhythmic drug therapy. The aim of the trial is to evaluate if the initial treatment choice (ablation vs. pharmacotherapy) influences AF disease progression, as measured by continuous cardiac monitoring. The outcomes of interest are disease progression, quality of life, and healthcare utilisation. The targeted population consists of healthy patients with symptomatic paroxysmal AF without clinically significant heart diseases aged between 18 and 75 years. This study represents a new research project leveraging the existing EARLY-AF randomised clinical trial infrastructure to examine the novel endpoints of: 1) disease progression ("time to first episode of persistent AF"), 2) progressive AF burden ("% time in AF"), 3) Quality of Life, and 4) healthcare utilisation at 36 months of follow-up.

DETAILED DESCRIPTION:
Project Aim: Atrial fibrillation is a major burden to healthcare systems. Contemporary costs of managing AF have been estimated to be up to 2.7% of total annual healthcare expenditures. A significant proportion of these expenses result from the direct costs associated with hospitalization and acute care. The CANet funded EARLY-AF Study aimed to determine whether EARLY invasive intervention resulted in a significant (i.e. >20%) reduction in arrhythmia recurrence and health care utilisation at one year of follow-up. The PROGRESSIVE AF study aims to evaluate the long-term effect of EARLY invasive intervention on disease progression and health care utilisation.

Project Background: Atrial fibrillation (AF) is a chronic progressive disease characterized by exacerbations and remissions. Early on, AF is triggered by one or more ectopic foci in the atria and is perpetuated via micro re-entrant circuits in the atrial body or at the pulmonary venous-left atrial junction. With recurrent episodes the atria undergoes electrical, contractile, and structural remodelling resulting in a greater predisposition toward sustained arrhythmia. This results in the progression of incidental and paroxysmal (self-terminating) AF to persistent (AF requiring intervention for termination) and eventually permanent AF (recurrent AF of >1 year in duration for which cardioversion was unsuccessful). While anti-arrhythmic drugs (AADs) remain the "first-line" therapy, these medications have only modest efficacy at maintaining sinus rhythm over the long term. Moreover, these agents are associated with significant non-cardiac side-effects (e.g. heart failure or organ toxicity), as well as the potential for pro-arrhythmia (i.e. increased propensity towards malignant arrhythmias). Conversely, multiple randomized controlled trials have demonstrated that catheter ablation is superior to drug therapy in maintaining sinus rhythm when AADs have been ineffective, are contra-indicated or cannot be tolerated.

While the evidence to date has demonstrated the universal superiority of ablation over AAD therapy, these studies have focused on medically refractory patients with more advanced forms of AF. While it has been postulated that early invasive intervention with catheter ablation may be beneficial, this assertion remains only hypothesis generating. As such we undertook the CANet funded EARLY-AF program. This multicenter collaboration sought to determine if an early invasive approach centered on cryoballoon based PVI was associated with a significant (i.e. >20%) reduction in arrhythmia episodes, AF symptoms, and healthcare utilization at one year of follow-up (i.e. the standard definition of success, as advocated by the Heart Rhythm Society).

In recent years attention has turned to longer-term effectiveness and safety outcomes, focusing more on the durability of catheter ablation procedures. Given that catheter ablation is being offered to relatively young and otherwise healthy patients as a first-line treatment approach, a comprehensive assessment of long-term clinical effectiveness is of particular importance with respect to informed decision-making. Moreover, a comprehensive understanding of the downstream effects of ablation greatly informs the evaluation of the cost-effectiveness of invasive AF ablation procedures.

The PROGRESSIVE AF project aims to leverage the infrastructure established with the EARLY-AF study to determine whether an a first-line invasive approach can alter the progressive pathoanatomical changes associated with AF, and by extension alter the disease trajectory (i.e. reduction in progression to persistent AF). The purpose of the current application is to undertake a 3 year follow-up study in order to better understand: 1) the natural history of AF (e.g. disease progression), 2) the relative ability of the two "first-line" treatment approaches to alter disease progression (e.g. AAD vs. pulmonary vein isolation), 3) the longer-term healthcare utilization associated with these two first-line treatment approaches, 4) the longer-term impact of these first-line approaches on patient reported outcomes.

Project Hypothesis, Research Question(s) and Objectives:

The majority of studies demonstrating the superiority of catheter ablation over anti-arrhythmic drug therapy have focused on medically refractory patients. This design pre-selects a group in whom medical therapy has been proven to be an ineffective therapy, and weights the benefit significantly towards the ablation arm. To date it is unknown whether the benefit of catheter ablation will be as substantial when delivered prior to medication failure (i.e. as a "first-line" ablation strategy). Moreover, it is unknown whether "first-line" ablation can alter the natural history of atrial fibrillation.

Project Hypothesis: We hypothesize that early intervention with the cryoballoon as a "first-line" therapy will favourably alter the natural history of AF when compared to an approach of "first-line" antiarrhythmic drug therapy. Specifically, we hypothesize that "first-line" ablation will result in increased freedom from recurrent arrhythmia, reduced need for pharmacologic or invasive intervention, reduced hospital utilisation due to symptoms caused by documented atrial arrhythmias, as well as a reduced progression from paroxysmal to persistent or permanent AF.

Objectives: The study is designed to evaluate of the impact of the early invasive management of AF with the Arctic Front cryoballoon. The primary objective of the study is to evaluate whether a "first-line" ablation strategy can reduce the progression from paroxysmal to persistent AF over ~36 months of follow-up, as detected by continuous cardiac monitoring. The secondary objective of the study is to evaluate the burden of AF on follow-up, as well as the health related quality of life (HRQOL) impact associated with early invasive intervention, in comparison to primary AAD therapy. This analysis will be centered on an evaluation of generic and disease-specific HRQOL instruments in order to determine the impact of an early invasive approach. The tertiary objective of the study is to evaluate the economic impact of early invasive intervention, with a focus on healthcare utilization. These will be used to derive a summary measure of health outcome and to inform subsequent healthcare resource allocation decisions.

ELIGIBILITY:
Inclusion Criteria:

* Non-permanent AF documented on a 12 lead ECG, Trans Telephonic Monitoring (TTM) or Holter monitor within the last 24 months
* Age of 18 years or older on the date of consent
* Candidate for ablation based on AF that is symptomatic
* Informed Consent

Exclusion Criteria:

* Regular (daily) use of a class 1 or 3 antiarrhythmic drug (pill-in-the-pocket AAD use is permitted) at sufficient therapeutic doses according to guidelines (flecainide >50 mg BID, sotalol >80 mg BID, propafenone >150 mg BID Previous left atrial (LA) ablation or LA surgery
* AF due to reversible cause (e.g. hyperthyroidism, cardiothoracic surgery)
* Active Intracardiac Thrombus
* Pre-existing pulmonary vein stenosis or PV stent
* Pre-existing hemidiaphragmatic paralysis
* Contraindication to anticoagulation or radiocontrast materials
* Left atrial anteroposterior diameter greater than 5.5 cm by transthoracic echocardiography
* Cardiac valve prosthesis
* Clinically significant (moderately-severe, or severe) mitral valve regurgitation or stenosis
* Myocardial infarction, PCI / PTCA, or coronary artery stenting during the 3-month period preceding the consent date
* Cardiac surgery during the three-month interval preceding the consent date
* Significant congenital heart defect (including atrial septal defects or PV abnormalities but not including PFO)
* NYHA class III or IV congestive heart failure
* Left ventricular ejection fraction (LVEF) less than 35%
* Hypertrophic cardiomyopathy (septal or posterior wall thickness >1.5 cm)
* Significant Chronic Kidney Disease (CKD - eGFR <30 µMol/L)
* Uncontrolled hyperthyroidism
* Cerebral ischemic event (strokes or TIAs) during the six-month interval preceding the consent date
* Pregnancy
* Life expectancy less than one (1) year
* Currently participating or anticipated to participate in any other clinical trial of a drug, device or biologic that has the potential to interfere with the results of this study
* Unwilling or unable to comply fully with study procedures and follow-up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of Persistent Atrial Tachyarrhythmia | Between 91 days following treatment initiation to final follow-up (~36 months)
  time to first occurrence of symptomatic or asymptomatic persistent atrial tachyarrhythmia (atrial fibrillation [AF], atrial flutter [AFL], or atrial tachycardia [AT]), as defined as the first occurrence of a continuous atrial tachyarrhythmia episode lasting ≥ 7 days in duration, or lasting 48 hours to 7 days in duration but requiring cardioversion for termination, as documented by implantable loop recorder.

SECONDARY OUTCOMES:
Atrial Fibrillation Burden | Treatment initiation to final follow-up (~36 months)
  Percentage time in atrial fibrillation
Health Related Quality of Life | Baseline, 12, 24, and 36 months following treatment initiation
  Change in disease-specific AFEQT score, and Generic EQ-5D score from baseline
Symptom Status | Baseline, 12, 24, and 36 months following treatment initiation
  Number of participants free from symptoms attributable to atrial fibrillation
Healthcare utilisation | Treatment initiation to final follow-up (~36 months)
  Number of participants experiencing an emergency department visit, cardioversion, and hospitalization >24 hours in a healthcare facility
Non-Protocol Ablation Procedure | Treatment initiation to final follow-up (~36 months)
  Number of patients experiencing a repeat ablation procedures in those randomized to first line catheter ablation, or any ablation procedure performed in patients randomized to AAD therapy
Safety Outcomes related to Ablation or AAD therapy | Treatment initiation to final follow-up (~36 months)
  Number of patients experiencing a major complication of ablation, or significant adverse drug events (death, ventricular pro-arrhythmia, syncope, hypotension, pacemaker insertion).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Andrade, Principal Investigator — Vancouver General Hospital
Locations (18):
- Canada (18):
  - Libin CV, Calgary, Alberta
  - Royal Alexandra, Edmonton, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - Vancouver General, Vancouver, British Columbia
  - Royal Jubillee, Victoria, British Columbia
  - QE II, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Mary's, Kitchener, Ontario
  - LHSC, London, Ontario
  - Southlake, Newmarket, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Rouge Valley, Scarborough Village, Ontario
  - St. Michael's, Toronto, Ontario
  - McGill, Montreal, Quebec
  - Sacre-Coeur, Montreal, Quebec
  - Laval, Québec, Quebec
  - CHUS Le Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - U Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided